CLINICAL TRIAL: NCT00657280
Title: Effect of Sitagliptin on Insulin Resistance and Myocardial Metabolism in Heart Failure
Brief Title: Study of the Effect of Sitagliptin on Glucose (Sugar) Metabolism in Patients With Heart Failure
Acronym: S-001
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael Fowler, PI, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04082008-1088
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects recieve Sitagliptin (Experimental): All subjects are aware of what they are taking. Nobody is blinded in this study. study
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — No one is blinded to the treatments.
  Other Names: Januvia

SUMMARY:
This study will investigate the effects of sitagliptin, a medicine commonly used to treat type 2 diabetes, on the utilization of glucose by the heart in patients with heart failure which is not due to heart attacks. We hope to determine whether improving the heart's ability to use glucose in the blood may help improve the function of the heart as well. If so, this may suggest that even people who do not have frank diabetes but who do have heart failure may benefit from using this medication.

This study will also investigate the effect of sitagliptin on the body's use of sugar, and of the effect of sitagliptin on blood flow to the heart.

DETAILED DESCRIPTION:
Screening:

Patients will be screened based on existing clinic information regarding NYHA class (New York Heart Association functional class) and heart failure characteristics. Patients will be approached in clinic after completing clinical care for that visit regarding participation in this trial.

If the patient agrees to participate, informed consent will be obtained at this time.

At enrollment:

Patients will be queried as to whether they have undergone previous nuclear medicine scans in the previous year in order to ensure that they do not exceed current standards for total annual radiation exposure.

Undergo a baseline combined 18-FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) PET/13N-NH3 PET/CT to assess the heart's ability to utilize blood sugar and coronary blood flow. This will take approximately 3-4 hours. This is a nuclear medicine procedure which is commonly used to assess myocardial viability as well as global heart function. It involves injection of a radioisotope-labeled tracers (18-FDG and 13N-NH3) intravenously followed by the measurement of myocardial uptake using a tomographic scanner. Venous blood samples performed during a 75g oral glucose load during the 18-FDG portion will assist with quantitation of myocardial glucose uptake and of measurements of insulin sensitivity. Perfusion (13N-NH3) images will be repeated during infusion of adenosine 0.14 mg/kg/min in order to assess coronary flow reserve. A computed tomography scan will be performed at the same time as the baseline PET scan for attenuation correction. Blood draws to measure changes in fasting insulin, blood sugar, lipid profile, and ADMA levels. Approximately 45 cc or 3 tablespoons of blood will be drawn and saved for possible future analysis.

18-FDG/13N-NH3 PET scans are routinely performed on patients with ischemic heart disease. While this study will use standard protocol for these examinations, they are not currently part of standard of care for nonischemic heart failure. However, they are important in testing the hypothesis of this study.

3) Begin sitagliptin 100 mg daily for four weeks. If calculated creatinine clearance is 30-49 cc/min by the Cockcroft-Gault formula, sitagliptin dose will be reduced to 50 mg daily for four weeks as per manufacturer guidelines. There will be no placebo arm. This will be an open-label study. Patients will be advised regarding potential side effects to prompt notification of study personnel. They will be instructed to contact the investigators for any concerns or evidence of adverse effects.

4) At four weeks: Repeat FDG/NH3 PET as above to compare to pretreatment scan. This will take approximately 3-4 hours. Blood draws to measure changes in fasting insulin, blood sugar, lipid profile, and ADMA (asymmetrical dimethylarginine) levels. Approximately 45 cc or 3 tablespoons of blood will be drawn and saved for possible future analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of nonischemic dilated cardiomyopathy, current NYHA class I-III congestive heart failure
2. Treatment with a stable comprehensive heart failure regimen for at least 3 months (including beta-blockers and ACE-inhibitors or angiotensin receptor blockers unless intolerant)
3. Age > 18 yrs

Exclusion Criteria:

1. Cardiomyopathy primarily due to one of the following:

   1. Ischemic heart disease
   2. Primary valvular lesion
   3. Hypertrophic cardiomyopathy
2. Cardiac resynchronization within the last 3 months
3. Calculated creatinine clearance <30 ml/min or end-stage renal disease on dialysis. Creatinine clearance will be determined by the Cockcroft-Gault formula.
4. Diagnosis of diabetes mellitus by:

   1. Diabetes previously diagnosed per patient history
   2. 2 or more fasting glucose values > 125 mg/dl
5. History of heart transplantation
6. Pregnancy or active breast feeding
7. Hospitalization for decompensated heart failure within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Fowler, Principal Investigator — Stanford University; Ronald M. Witteles MD, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: There is only one group. All the participants took Sitagliptin 100mg daily and acted as their own controls
Period: Overall Study
Arm/Group | Sitagliptin
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult patients diagnosis of nonischemic dilated cardiomyopathy with Class I-III symptoms. all patients were required to have been on a stable comprehensive heart failure regimen for at least three months, including therapy with beta-blockers and angiotensin-converting-enzyme inhibitors or angiotensin-receptor-blockers unless they were intolerant.
Groups:
- Sitagliptin: There is only one group. All the participants took the Sitagliptin.
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 51 [43 to 60]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Effects of Sitagliptin on Myocardial Glucose Uptake Measured by Myocardial PET Scan
Description: This study will investigate the effects of sitagliptin, a medicine commonly used to treat type 2 diabetes, on the utilization of glucose by the heart in patients with heart failure which is not due to heart attacks. We hope to determine whether improving the heart's ability to use glucose in the blood may help improve the function of the heart as well. If so, this may suggest that even people who do not have frank diabetes but who do have heart failure may benefit from using this medication. Baseline glucose uptake scans will be compared with the scans on sitagliptin thirty days after baseline
Time Frame: 30 days
Population: Scans were lost in 4 participants
Measure: Mean (Full Range); unit: SUV
Arm/Group | Sitagliptin
Number analyzed (Participants) | 12
SUV
  Baseline | 3.4 [2 to 6]
  30 days | 4.1 [3 to 6]

2. Primary Outcome: Determine the Effects of Sitagliptin on Myocardial Glucose Uptake in Patients With Nonischemic Cardiomyopathy
Description: This study will investigate the effects of sitagliptin, a medicine commonly used to treat type 2 diabetes, on the utilization of glucose by the heart in patients with heart failure which is not due to heart attacks. We hope to determine whether improving the heart's ability to use glucose in the blood may help improve the function of the heart as well. If so, this may suggest that even people who do not have frank diabetes but who do have heart failure may benefit from using this medication.
Time Frame: 2008-2012
Reporting Status: Not Posted

3. Secondary Outcome: Determine the Effects of Sitagliptin on Microvascular Function in Patients With Nonischemic Cardiomyopathy
Time Frame: 2010-2012
Reporting Status: Not Posted

4. Secondary Outcome: Determine the Effects of Sitagliptin on Microvascular Function in Patients With Nonischemic Cardiomyopathy
Description: as for outcome 2
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No